CLINICAL TRIAL: NCT01803061
Title: Use of Computer-based Patient-reported Data to Assess Long Term and Late Effects of Head and Neck Cancer at the Point-of-care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Cancer Society (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); Sygekassernes Helsefond (Other)
Responsible Party: Principal Investigator, Trille Kjær, Phd student, Danish Cancer Society
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WebCan
Record Dates: First submitted 2013-02-21; First posted 2013-03-04 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Head and Neck Cancer Patients; Late Effects
Keywords: Head and neck cancer; Quality of life; Symptom-burden; Late effects
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WebCan (Experimental): Provides computerized PRO to the treating physician at the point of care
  Interventions: Behavioral: WebCan
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: WebCan — Provide computerized PRO (Patient Reported Outcome) to treating physician at the point of care to assess late effects after head and neck cancer
  Arms: WebCan

SUMMARY:
Patient-reported information on outcomes such as symptom-burden and health-related quality of life (QoL) is regarded as a useful tool to improve quality of care in clinical cancer research. However, integrating patient-reported information in the routine clinical practice is often difficult due to excessive time use and practical barriers. Electronic data acquisitions, where the treating physician has immediately access to the patient-reported data in the subsequent consultation, have been shown to be beneficial in the everyday clinical decision making.

The aim of this study is to develop and test a computer-based patient-reported assessment tool that will assist the clinicians in tracking long term and late effects in head and neck cancer patients and investigate if the tool leads to improved symptom assessment of a range of head and neck cancer specific symptoms, which again may lead to improved symptom control and enhanced quality of life in the patients.

Patients with a diagnosis of head and neck cancer attending the oncology outpatient clinics at Herlev Hospital and physicians and nurses who work at the clinic will be invited to participate. The assessment tool will be developed with inspiration from prior international studies of symptom assessment in head and neck cancer patients and tailored so that it will fit into a Danish context. The tool will be tested in a controlled intervention study. In the intervention group, patients will complete the assessment tool in the patients waiting area prior to every scheduled consultation. The result will then be printed and provided to the treating physician. In the control group, the patients will complete the assessment tool prior to consultations. However, the data will not be provided to the physicians at any time.

To assess the impact of the tool on number of symptoms addressed during consultations and patients' overall quality of life, medical records will be reviewed for before start of intervention and again at 6 and 12 months follow-up. The patients will also complete the EORTC QLQ-C30 and the EORTC QLQ-H&N35 at baseline and at 6 and 12 months follow-up. Furthermore, we will conduct a qualitative evaluation (semi structured interview and participant observations) of attitudes among clinicians and patients regarding the use of tool at the point of care.

ELIGIBILITY:
Inclusion Criteria:

* Prevalent recurrence free patients with cancers in the tongue, oral cavity, pharynx and larynx attending the oncology clinic at Herlev Hospital, Herlev, Denmark. 9 months to 5 years after end of treatment

Exclusion Criteria:

* Patients with recurrence of their cancers and patients still in treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of late effects | baseline, 6 and 12 months follow-up

SECONDARY OUTCOMES:
Quality of life | baseline, 6 and 12 months follow-up
  Quality of life at baseline and 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Johansen, Professor, Study Director — Danish Cancer Society Research Center
Locations (2):
- Denmark (2):
  - Herlev Hospital, Herlev
  - Danish Cancer Society Research Center, Unit of Suvivorship, Copenhagen, Ø